CLINICAL TRIAL: NCT03092986
Title: Outcome of Cisplatin and Vinblastine Versus Paclitaxel and Carboplatin as Sequential Chemotherapy Followed by Radiotherapy in Locally Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Anshu Kumar Thakur, MD Oncology program Phase B Resident Doctor,Department of Oncology,Principal investigator., Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BangabandhuONCOLOGY
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Vinblastine; Radiotherapy, Conformal

STUDY DESIGN:
Intervention Model Description: Randomized Controlled type, 60 patients randomized with help of randomized number generator in two arms, Arm A and Arm B, each with at least 30 number of patients, research material will be data collection form,Arm A will receive paclitaxel 200 mg/m2 i.v over 3 hrs on D1; carboplatin AUC 6 i.v over 60 minutes on D1 every 3 wks for 2 cycles followed by radiotherapy with 6000 c Gy given in 30 fractions beginning on day 42 , Arm B willl receive - cisplatin (100 mg/m2 BSA i.v over 2 hrs. on days 1 and 29) and vinblastine (5 mg/m2 BSA i.v rapidly push weekly on days 1,8,15,22 and 29) followed by radiotherapy with 6000 cGy given in 30 fractions beginning on day 50 ,data will be analysed and interpreted and result will be drawn on basis of outcome measures which is again based on tumor response RECIST criteria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- chemotherapy with paclitaxel and carboplatin (Active Comparator): Intervention: paclitaxel 200 mg/m2 AUC and carboplatin AUC 6 on day 1 every 3 wks for 2 cycles followed by three dimensional conformal radiotherapy on day 42
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: three dimensional conformal radiotherapy
- chemotherapy with cisplatin and vinblastine (Experimental): Intervention : cisplatin 100 mg/m2 on day 1 and 29 and vinblastine 5mg/m2 on days 1,8,15,22 and 29 followed by three dimensional conformal radiotherapy on day 50
  Interventions: Drug: Cisplatin; Drug: Vinblastine Sulfate; Radiation: three dimensional conformal radiotherapy

INTERVENTIONS:
Drug: Paclitaxel — paclitaxel 200 mg/m2 i.v over 3 hrs on day 1, every 21 days for 2 cycles followed by radiotherapy on day 42
  Other Names: Xelpac
  Arms: chemotherapy with paclitaxel and carboplatin
Drug: Carboplatin — carboplatin AUC 6 iv over 1 hr on day 1 , every 212 days for 2 cycle followed by radiotherapy on day 42
  Other Names: carboplat
  Arms: chemotherapy with paclitaxel and carboplatin
Drug: Cisplatin — cisplatin 100 mg/m2 i.v over 2 hrs on day 1 and 29 followed by radiotherapy on day 50
  Other Names: Platinex
  Arms: chemotherapy with cisplatin and vinblastine
Drug: Vinblastine Sulfate — Vinblastin 5mg/m2 i.v on day 1,8,15,22 and 29 followed by radiotherapy on day 50
  Other Names: Velvin
  Arms: chemotherapy with cisplatin and vinblastine
Radiation: three dimensional conformal radiotherapy — three dimensional conformal radiotherapy would be given at day 42 after completion of paclitaxel and carboplatin 2 cycle and at day 50 after completion of cisplatin and vinblastin from d1 to d29

SUMMARY:
Lung cancer is the leading malignancy worldwide and in Bangladesh. Most of the lung cancer is of Non-small Cell Lung Cancer (NSCLC) type. For locally advanced NSCLC, combined modality treatment is required. Concurrent chemo-radiotherapy and sequential chemo-radiotherapy are the two recommended options. Sequential chemo-radiotherapy is mainly practiced in Bangladesh due to its less toxicity profile. There is no head to head comparative study done which focuses on the sequential chemotherapy regimens used in locally advanced NSCLC.

Hypothesis:

Null Hypothesis (H0): Sequential chemotherapy with cisplatin and vinblastine followed by radiotherapy and paclitaxel and carboplatin followed by the same radiotherapy in locally advanced NSCLC, there is no difference in loco-regional tumor control.

Alternative Hypothesis (HA): Sequential chemotherapy with cisplatin and vinblastine followed by radiotherapy and paclitaxel and carboplatin followed by the same radiotherapy in locally advanced NSCLC, cisplatin and vinblastine is more responsive and effective in loco-regional tumor control than paclitaxel and carboplatin.

DETAILED DESCRIPTION:
Lung cancer is the leading malignancy worldwide and in Bangladesh. Most of the lung cancer is of Non-small Cell Lung Cancer (NSCLC) type. For locally advanced NSCLC, combined modality treatment is required. Concurrent chemo-radiotherapy and sequential chemo-radiotherapy are the two recommended options. Sequential chemo-radiotherapy is mainly practiced in Bangladesh due to its less toxicity profile. There is no head to head comparative study done which focuses on the sequential chemotherapy regimens used in locally advanced NSCLC.

Aim and Objective:

To compare treatment outcome and acute toxicities between two standard sequential chemotherapy regimens (Cisplatin and Vinblastine followed by radiotherapy and Paclitaxel and Carboplatin followed by same radiotherapy) in patients with locally advanced stage III NSCLC.

Material and Method:

A total number of 60 patients, who are clinically locally advanced (stage III A and III B), histologically proven NSCLC, inoperable and with ECOG performance score upto grade 2 and body weight loss <10 % in 3 months will be included in this study.

Patients will be randomly assigned to receive either Arm A or Arm B. Arm A will receive - paclitaxel 200 mg/m2 body surface area(BSA) i.v over 3 hrs on D1; carboplatin Area Under Curve(AUC) 6 i.v over 60 minutes on D1 every 3 wks for 2 cycles followed by radiotherapy with 6000 (Centigray)c Gy given in 30 fractions beginning on day 42 And Arm B will receive - cisplatin (100 mg/m2 BSA i.v over 2 hrs. on days 1 and 29) and vinblastine (5 mg/m2 BSA i.v rapidly push weekly on days 1,8,15,22 and 29) followed by radiotherapy with 6000 cGy given in 30 fractions beginning on day 50 .

All patients will be followed up as per guideline for 6 months in this study. Discussion: All the relevant data will be compiled on a master chart first and then statistical analysis of the results will be obtained by using Window based computer software devised with Statistical Packages for Social Sciences (SPSS-17) (SPSS Inc, Chicago Illinois(IL) USA). The data will be analyzed using Chi-square test and 'T' test and association will be analyzed by Pearson's correlation coefficient (r value) test. The results will be presented in tables, figures, diagrams. Significant value of 'p' will be decided at a level of 0.05 in two tailed tests.

Selection of patients:

A. Inclusion Criteria:

* Patients with locally advanced (stage III a, b) NSCLC.
* Patients who are inoperable. Patients Eastern Co-operative Group (ECOG) performance score up to grade 2.

B. Exclusion Criteria:

* Age below 18 years.
* Patients with history of prior chemotherapy or radiotherapy to lung region.
* Serious concomitant medical illness including severe heart disease, uncontrolled diabetes mellitus or hypertension.
* Life expectancy < 6 months.
* Patient with uncontrolled infection
* Pregnant or lactating woman.
* Psychiatric illness.

Minimum laboratory criteria required to include:

* Hemoglobin should be more than 10 gm. /dl or more than 60%.
* An absolute white blood count(WBC) more than or equal to 4000 cells/mm3.
* Platelet count more than or equal to 100000 cells/mm3.
* Bilirubin level should be equal to or less than 1.5 mg/dl.
* SGPT(serum glutamic-pyruvic transaminase) level not more than 4 times of the upper limit.
* Serum creatinine level should be equal to or less than 1.5 mg/dl.
* Blood Urea level less than 50 mg/dl. Sampling technique Randomized number generator, a random number generator is a computational process that produces random numbers by using statistical algorithm.

Outcome measures:

table- clinical response , a 3rd follow up at week 30 after completion of treatment for both the arms (n=60)

response Arm A Arm B X2 value P value Complete response (CR) Partial response (PR) Progressive disease (PD) Stable disease (SD)

Responses Description Complete Response ( CR ) Disappearance of all known diseases, confirmed at ≥ 4 weeks Partial Response ( PR ) ≥ 50 % decrease from baseline, confirmed at ≥ 4 weeks.

Progressive disease ( PD ) ≥ 25 % increase in one or more lesions or appearance of new lesions Stable disease ( SD ) Neither PR or PD criteria met

ELIGIBILITY:
Inclusion Criteria:

* • Patients with locally advanced (stage III a, b) non-small cell lung cancer.

  * Patients who are inoperable. Patients Eastern Co-operative Group (ECOG) performance score up to grade 2.

Exclusion Criteria:

* • Age below 18 years.

  * Patients with history of prior chemotherapy or radiotherapy to lung region.
  * Serious concomitant medical illness including severe heart disease, uncontrolled diabetes mellitus or hypertension.
  * Life expectancy < 6 months.
  * Patient with uncontrolled infection
  * Pregnant or lactating woman.
  * Psychiatric illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
tumor response | 30 weeks
  complete response(CR), partial response(PR), progressive disease(PD) and stable disease(SD),Responses Description Complete Response ( CR ) Disappearance of all known diseases, confirmed at ≥ 4 weeks.
  Partial Response ( PR ) ≥ 50 % decrease from baseline, confirmed at ≥ 4 weeks. Progressive disease ( PD ) ≥ 25 % increase in one or more lesions or appearance of new lesions Stable disease ( SD ) Neither PR or PD criteria met final tumor response will be seen in 30 weeks of starting of completion and will be considered as the primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology,Bangabandhu Sheikh Mujib Medical university, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No